CLINICAL TRIAL: NCT06855017
Title: Writing: a Factor That Can Influence Understanding of Prescriptions in the Geriatric Population
Acronym: ROSA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240298; 2024-A00580-47 (Other: IDRCB)
Record Dates: First submitted 2025-02-20; First posted 2025-03-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prescription Medication Understanding
Keywords: geriatry; prescription medication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients over 75
  Interventions: Other: create a pillbox day

INTERVENTIONS:
Other: create a pillbox day — create a pillbox day based on two separate fictitious prescriptions

SUMMARY:
Understanding prescriptions is a key factor in the therapeutic education and compliance of elderly patients with multiple medications. However, the way prescriptions are written and typed depends on doctors' habits, due to a lack of recommendations on the subject.

The introduction of a state-qualified nurse to manage treatment will soon be a public health issue, given the ageing population and human resources problems.

The hypothesis is that certain editorial and typographical choices can make prescriptions clearer, and could thus help elderly patients, either cognitively unaffected or at risk of cognitive fragility, to better understand their prescriptions and thus limit the risk of medication errors.

DETAILED DESCRIPTION:
Patients over 75 years of age represent the largest group of drug users. This is also the group with the highest risk of medication-use errors. These elderly, polymedicated people are subject to frequent changes in treatment, particularly when discharged from hospital, where on average 2 out of 3 prescriptions are changed, with more than 6 changes per prescription. Furthermore, up to 75% of the elderly are unable to provide details of their prescriptions, and almost half misinterpret them.

These data are indicative of poor compliance in geriatrics. Compliance is defined as the degree of concordance between an individual's behavior and medical prescriptions or recommendations. The factors contributing to poor compliance in elderly patients have been studied in numerous studies. The following 4 categories of factors have been identified:

* The first category corresponds to the treatments themselves: unsuitable galenic form, difficult-to-obtain dosage, misunderstood mode of administration, similar packaging and tablets, handling of eye drops, liquids to be measured, blister pack openings, handling of pillbox, size of tablets to be handled (too small) or swallowed (too big), poor tolerance.
* The second category corresponds to patients' comorbidities, including cognitive and functional deficits (dexterity, vision), depressive or anxious state, as well as patients' level of literacy, defined as the ability to read, understand and use written information in daily life, and numeracy, defined as the fundamental mathematical knowledge enabling a person to function in society.
* The third category relates to the disease: the patient's own representations and perceptions of the disease, as well as his or her habits.
* The fourth category relates to the relationship between doctor and patient: clarity of repeated explanations given to the patient, empathy, partner relationship, patient not daring to express problems of understanding.

In addition to all these factors limiting compliance, the investigator hypothesized that poor understanding of prescriptions could lead to poor patient compliance and medication errors.

In fact, it's common to complain about doctors' handwriting and the resulting lack of understanding of prescriptions. But we believe that beyond the practitioner's handwriting, all the editorial and typographical elements of the prescription come into play in its comprehensibility.

There is no reference or recommendation on how to mention the various elements on a prescription. Practitioners are free to make the editorial and typographical choices they wish. The investigator define the editorial quality of a prescription as the art of writing down instructions designed to facilitate reading, such as the choice of typeface, font size, spacing and the absence of abbreviations.

The interest in studying a geriatric population more specifically is to look at the specific impact of frailty in relation to aging on the understanding of the prescription, in order to better understand its elements. Frailty is defined by the presence of geriatric syndromes such as neurocognitive disorders, mood disorders, undernutrition and gait disorders. Geriatric syndromes are systematically identified during hospitalization as part of the standardized geriatric assessment.

Physiological aging can be defined as a reduction in reserves. Cognitive physiological aging is thus marked by a decline in attention, working memory and executive functions. These are the processes involved in making a pillbox. As a result, an elderly person with no neurocognitive problems will have more difficulty completing a pillbox than a younger person.

Pillboxing is even more difficult in patients with neurocognitive disorders. We are only interested in patients with a mild neurological disorder, i.e., according to the Diagnostic and Statistical Manual -5 (DSM-5), presenting an acquired, significant and progressive reduction in ability in one or more cognitive domains, but with preserved autonomy to perform simple activities of daily living. In these patients, complex instrumental activities of daily living (such as paying bills or managing medication intake) are preserved, but greater effort, compensatory strategies or accommodation may be required.

The aim of this study is to determine what editorial and typographical choices could be made to increase patient understanding of prescriptions, with a view to improving physician practice. To this end, eligible patients will be asked to create a day's pillbox from prescriptions with varying wording and typographical choices. The investigators also want to show that a common practice in prescription writing, although normally prohibited by law, is to use the trade name for frequent medications without mentioning the INN, which can lead to errors in patients' medication use.

Each eligible patient will be asked to create a pillbox day based on two separate fictitious prescriptions. Each of the two prescriptions will consist of 7 prescription lines. The first prescription line of the first prescription will be equivalent to the first prescription line of the second prescription in terms of the number of tablets/capsules to be taken and the frequency during the day, and so on for the 7 prescription lines, but the editorial and typographical choices will be different. One of the two prescriptions will comply with the legislation, and will present the editorial and typographical choices which, according to the literature, would promote comprehension. We'll call this prescription the optimized prescription. This prescription will be similar for all patients, except for the names of the active ingredients. For each prescription line, two active ingredients are possible, and a draw will decide which active ingredient will be the one on the optimized prescription and which will be the one on the other prescription. On the other prescription, which we'll call the test prescription, each possible editorial and typographical choice will be drawn at random to appear or not.

In short, each eligible patient will successively read two prescriptions: the optimized prescription, which will be similar for each participant (except for the names of the active ingredients), and the test prescription, which will vary for each patient. Each patient will thus be his or her own witness. The order in which each of the two prescriptions is read will be drawn at random for each patient, to limit learning bias or, on the contrary, fatigue.

To set up the two prescriptions, we established a number of possible choices, based on the literature and guides such as Unapei's "Facile à Lire et à Comprendre" and "Santé pour Tous en pays Breton".

We selected 13 different editorial and typographical variations to test with our study. The editorial variations selected for the study are as follows:

* The use of abbreviations or not,
* Writing 0.5 or 1/2 or a half *,
* Writing the number of tablets/capsules as a letter or a number,
* Write with or without particularization. Particularization means linking each tablet to a specific time of intake (morning, noon and evening). This avoids inferences. An inference is a logical operation of deduction/reasoning to make explicit information that is only evoked or assumed to be known,
* Write the rhythm as "3/J" without precision, to mean "morning, noon and evening*".
* Choose to write the dosage in metric units of mass (which may require the patient to calculate the number of tablets/capsule required) or in number of tablets/capsule.
* Write the brand name or INN of a treatment (this is a matter of legislation and not a simple editorial choice). We have chosen the case of amoxicillin-clavulanic acid, often prescribed under the name Augmentin on prescriptions*.

  * The 3 variations marked with an asterisk above are presumed to be particularly confusing and will be given special treatment during randomization and analysis.

The typographical variations selected are as follows:

* Italicized or not,
* Bold or not,
* Writing in upper or lower case,
* Writing in a serif font (Times New Roman) or sans serif font (Arial),
* Font size 10 or 12,
* Write with or without line feed.

On the optimized prescription, there are no abbreviations, half a tablet is written in full, the number of tablets/capsule is written in Arabic numerals, each tablet is linked to a precise time of intake, there are no calculations to be made to determine dosage, the name of the active ingredient is written in INN, there are no italics, no bold, no capitals, the font is sans serif, the font size is 12 and there is a line break between each treatment.

Conversely, on the test prescription, the 10 variations not marked with an asterisk may or may not appear, depending on the draw (a different draw for each of these 10 possible variations). For the remaining 3 variations, they appear systematically on the test prescription, without random selection, each on a single line: the use of the "3/J" formulation, the writing of "0.5" or "1/2" instead of "half", and the use of "Augmentin" instead of "Amoxicillin clavulanic acid" (these variations seem particularly confounding and could overwhelm the effect of the others in a factorial experimental design).

For the editorial variations whose presence on the test prescription is randomly selected, of which there are four, there is (i) the use of abbreviations ("cp/gl" instead of "tablet/capsule"), (ii) the writing of capsule/tablet numbers in figures, (iiii) an absence of particularization and (iv) dosage written using the metric system, these variations then appear on all prescription lines.

For typographical variations, of which there are six, the typography can be with a serif font, in uppercase, bold, italic, without line break, and these variations also appear on all prescription lines.

Finally, here is the list of drugs drawn at random for each of the 7 prescription lines (randomly one will be on the optimized prescription, the other on the test prescription):

* Line 1: Diffu K 200 mg or Paracetamol 500 mg
* Line 2: Seresta 10 mg or Prednisolone 5 mg
* Line 3: Fumafer 66 mg or Folic Acid 5 mg
* Line 4: Mianserin 10 mg or Temesta 1 mg
* Line 5: Phloroglucinol 80 mg or Levothyroxine sodium 25 µg
* Line 6: Amoxicillin-clavulanic acid for optimized prescription and Augmentin for test prescription
* Line 7: Furosemide 40 mg or Bisoprolol 2.5 mg

In a second phase, the analysis will determine which factors (age, gender, socio-educational level, co-morbidities including neurocognitive disorders, geriatric syndromes) have the greatest influence on prescription comprehension.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following criteria may be included in the study:

* Patients over 75 years of age,
* hospitalized in the UGA and/or SMR at Bretonneau, apart from a still active acute/confusional episode
* Presenting a cognitive assessment by MMSE greater than or equal to 20
* accustomed to making their own pill dispenser at home, with the presence of a state-qualified nurse for other tasks (dressing/compression stockings/controls, etc.) not excluded -

Exclusion Criteria:

Patients with the following criteria cannot be included in the study:

* Obvious sensory disorders, at the discretion of the physician:

  * Disabling hearing problems without hearing aids, preventing them from following a conversation
  * Visual impairment preventing reading
* Dexterity problems preventing the handling of medication blisters (e.g. stroke with severe motor impairment of the right upper limb, uncontrolled Parkinson's disease, etc.).
* Poor command of the French language/illiteracy
* Patients under guardianship or curators
* No affiliation to a social security scheme
* Patient under AME
* Opposition to participation in research

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Any patient aged over 75, male or female, hospitalized at Bretonneau in an Acute Geriatric Unit (UGA) or in Medical and Rehabilitation Care (SMR), other than in the event of a persistent acute episode or confusion, who previously managed his or her treatments at home using a pillbox, and who has an MMSE of over 20 (a test performed systematically as part of the department's standardized geriatric assessment), is eligible.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
number of errors made by the patient included when creating a day's pillbox based on the optimized prescription | 1 day
number of errors made by the patient included when creating a day's pillbox from the test prescription | 1 day

SECONDARY OUTCOMES:
Number of pillbox errors when the patient is exposed to abbreviations | 1 day
Number of errors when the patient is exposed to a number of capsules/tablets written in figures rather than in words | 1 day
Number of errors when the patient is exposed to an unspecified intake rhythm | 1 day
Number of errors when the patient is exposed to a mass dosage rather than a number of tablets/capsules | 1 day
Number of errors when the prescription is in italics | 1 day
Number of errors when the prescription is in bold | 1 day
Number of errors when the prescription is in upper case | 1 day
Number of errors when the prescription is in Times New Roman with serif | 1 day
Number of errors when the prescription is in size is 10 | 1 day
Number of errors when the prescription is in Arial, without serif | 1 day
Number of errors when the order does not space its lines | 1 day
Proportion of patients making an error on amoxicillin-clavulanic acid when written as "Augmentin". | 1 day
Proportion of patients making an error on a prescription line with a "3/D" dosing interval | 1 day
Proportion of patients making an error on the prescription line containing the wording "0.5" or "1/2" (drawn randomly) instead of "one half" | 1 day
pillbox creation time from test prescription (all variations aggregated) | 1 day
time to create a pillbox from a optimized prescription | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Golstein, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Bretonneau, Paris, France